CLINICAL TRIAL: NCT00727922
Title: Evaluation of Mangafodipir Protective Activity Against Oxaliplatin Neurotoxicity
Brief Title: Protective Effect of Mangafodipir Against Oxaliplatin Neurotoxicity
Acronym: MnDPDP-K04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P071203
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Neurotoxic Disorders; Cancer
Keywords: Neuropathy; Oxaliplatin; Mangafodipir
MeSH Terms: conditions — Neurotoxicity Syndromes; Neoplasms | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Mangafodipir

INTERVENTIONS:
Drug: Mangafodipir — Mangafodipir (0.5 ml/kg) is administered as a 30 minutes infusion just after each administration of oxaliplatin. The oxaliplatin dose (85 to 100 mg/m²) and the length of the infusion (2 hours) are the same that before the inclusion and modifications are not authorized during all the study participation. During 4 months (8 administrations).

SUMMARY:
Oxaliplatin is a major antitumor agent but its use is limited by potentially disabling neurotoxicity, characterized by a sensitive defect in the extremities.Mangafodipir is a MRI contrast agent with antioxidant properties. Our previous laboratory works showed that mangafodipir is able to prevent hematologic toxicity of several chemotherapy agents, including oxaliplatin and to increase their antitumor activity. Preliminary clinical data suggested that mangafodipir could prevent oxaliplatin neurotoxicity.The primary purpose of the present study is to assess the protective effect of mangafodipir in patients who have a already moderate oxaliplatin neuropathy and in whom the continuation of this treatment is desirable because of significant antitumor effect.

DETAILED DESCRIPTION:
Phase 2 study aiming to assess the protective effect of mangafodipir against the oxaliplatine neuropathy.Population: Cancer patient who have a mild (grade 2) oxaliplatin neuropathy and in whom the continuation of oxaliplatin for at least 4 infusions is desirable will be include, whatever the location of the primitive tumor and the use of others anticancer agents.Treatment: Mangafodipir (0.5 ml/kg) is administered as a 30 minutes infusion just after each administration of oxaliplatin. The oxaliplatin dose (85 to 100 mg/m²) and the length of the infusion (2 hours) are the same that before the inclusion and modifications are not authorized during all the study participation. Primary objective: Neuropathy are clinically evaluated according to NCI-CTC criteria before each mangafodipir and oxaliplatin and thereafter one month after the last infusion. The primary criteria is the worst grade of oxaliplatin neuropathy experienced by each patient. The improvement of neuropathy is defined as a decrease by at least one grade of the severity of the neuropathy for at least 2 months.

Hypothesis: at least 50% of patients will experience an improvement or a stabilization of the oxaliplatin neuropathy while receiving the mangafodipir - oxaliplatin association.Treatment discontinuation: the treatment will be stopped if the neuropathy worsened by at least one grade, in case of tumor progression, intolerable toxicity, and patient wish.

Number of patients: it will be determined according to a simplified Gehan procedure: The inclusions will be stopped if no objective response (neuropathy improvement) is observed among the first 9 evaluable patients. If at least one response is observed, 16 more evaluable patients will be include. The total number of patients will be between 9 and 30 patients, including non evaluable patients.

Pharmacokinetic: Serum and intra- erythrocytes manganese concentration will be evaluated before each mangafodipir infusion in order to detect accumulation Pharmacodynamic: plasmatic total antioxidant activity, superoxide dismutase activity and lipid peroxidation will be assessed at the first cycle: before and after the administration of oxaliplatin and just after the perfusion of mangafodipir.

ELIGIBILITY:
Inclusion Criteria:

* NCI CTC grade 2 or more neuropathy induced by oxaliplatine
* At least 18 years old
* ECOG PS: 2 or less
* Life expectancy longer than 3 months
* Written informed consent
* Adequate hematologic, liver and renal functions

Exclusion Criteria:

* Known hypersensibility to oxaliplatine
* Cancer resistant to oxaliplatine
* Fertile woman or man not willing to use adequate contraception
* Pregnant or lactating women
* Vitamin B6 administration within 48h prior to mangafodipir administration
* Uncontrolled infection
* Treatment with any other investigational agent, or participation in another clinical trial within 3 weeks prior to first administration of mangafodipir
* Evidence of any other disease or condition that contra-indicates the use of an investigational drug
* No Social Security insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Maximal neuropathy severity (NCI-CTC score) established before each oxaliplatin injection | every 15 days

SECONDARY OUTCOMES:
Number of oxaliplatin administration | every 15 days
Progression free survival (time from inclusion to cancer progression) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Alexandre, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Cochin, Paris, France

REFERENCES:
- [Result] Coriat R, Alexandre J, Nicco C, Quinquis L, Benoit E, Chereau C, Lemarechal H, Mir O, Borderie D, Treluyer JM, Weill B, Coste J, Goldwasser F, Batteux F. Treatment of oxaliplatin-induced peripheral neuropathy by intravenous mangafodipir. J Clin Invest. 2014 Jan;124(1):262-72. doi: 10.1172/JCI68730. Epub 2013 Dec 20. PMID 24355920